CLINICAL TRIAL: NCT06230887
Title: Implementation of Innovative Treatment for Moral Injury Syndrome: A Hybrid Type 2 Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Central Alabama Health Care System (Unknown); VA Atlanta Healthcare System (Unknown); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 22-132
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Moral Injury Syndrome
Keywords: Moral Injury; Posttraumatic Stress Disorder; Spirituality; chaplains
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the experimental condition (Building Spiritual Strength, an evidence-based, manualized, spiritually integrated group counseling program for moral injury/spiritual distress/values related distress associated with trauma) or the control condition (Present Centered Group Therapy, an evidence-based, manualized group treatment for PTSD.)
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not have access to shared files, and will not be at any team meetings in which individual participants are discussed, so she will not know to what condition the participants have been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Building Spiritual Strength (Experimental): Spiritually integrated group intervention for moral injury.
  Interventions: Behavioral: Building Spiritual Strength
- Present Centered Group Therapy (Active Comparator): Coping strategies group intervention addressing broad spectrum trauma symptoms
  Interventions: Behavioral: Present Centered Group Therapy

INTERVENTIONS:
Behavioral: Building Spiritual Strength — Spiritually Integrated group intervention for moral injury
  Arms: Building Spiritual Strength
Behavioral: Present Centered Group Therapy — Active control, manualized evidence-based coping skills intervention for PTSD
  Arms: Present Centered Group Therapy

SUMMARY:
Moral Injury Syndrome (MIS) affects up to 35-60% of Veterans managing combat-related PTSD; it results from experiences that challenge deeply held values or spiritual beliefs. Symptoms of MIS may include hopelessness, helplessness, loss of spiritual beliefs, difficulty with forgiveness, loss of meaning or purpose, reduced trust in self or others, or intractable guilt, shame or anger.

Veterans managing MIS have difficulty responding to mental health treatment, and are at increased risk for suicide ideation or attempts. To date evidence-based interventions for MIS are not widely available in VA. This study will implement an evidence-based intervention for MIS in four VA facilities, collect data on the effectiveness of the intervention, and develop an implementation toolkit. This data will inform national dissemination in collaboration with the Office of Mental Health and Suicide Prevention and the National Chaplain Service.

DETAILED DESCRIPTION:
Background: Moral injury syndrome (MIS) consists of the psychological and behavioral sequelae of experiences that challenge moral, spiritual, or values related beliefs. Symptoms of MIS may include hopelessness, helplessness, loss of previously held spiritual beliefs, struggle with a Higher Power, difficulty with forgiveness, lack of meaning or purpose, reduced trust in self or others, or intractable guilt, shame or anger. Individuals managing MIS are up to twice as likely as their peers to consider and attempt suicide, and derive less benefit from psychotherapy. There are few evidence-based interventions for moral injury; one such intervention is a manualized, group intervention called "Building Spiritual Strength (BSS)." In previous randomized controlled trials BSS has been shown to reduce both symptoms of PTSD and spiritual distress.

This clinical trial will be one of the first to measure symptoms of MIS as a primary outcome. Hypotheses are:

1. Compared to Present Centered Group Therapy (PCGT), BSS will significantly decrease symptoms of MIS.
2. Compared to PCGT, BSS will significantly decrease symptoms of PTSD, depression, and suicidal ideation.

Significance: To date there are not standard procedures for assessing and treating MIS, so it is likely that untreated MIS is contributing to poor outcomes, including suicides. Developing an implementation toolkit so that BSS is widely available in VA facilities could reduce the impact of MIS on Veterans' mental health.

Innovation and Impact: To date there have not been funded implementation studies on treatments for MIS in Veterans, and very few VA facilities provide evidence-based care for MIS. This study can clear the way to make evidence-based care for MIS more accessible in the VA system.

Specific Aims:

1. Conduct a mixed methods pre-implementation evaluation to identify barriers and facilitators for BSS implementation at each site, and to develop local implementation strategies. Specific implementation variables assessed, based on the Proctor and EBQI models include acceptability, appropriateness, and feasibility. Specific variables to be assessed will include a) acceptability of BSS to stakeholders, b) available implementation resources, and c) organizational openness to adding a new EBP.
2. Conduct a randomized controlled trial comparing BSS to Present Centered Group Therapy (PCGT) for Veterans who score above cutoff on the Moral Injury Outcomes Scale. Effectiveness and functional outcomes will be informed by the psychospiritual developmental model of MIS.
3. Conduct a mixed methods post-implementation evaluation to compare outcomes across chaplaincy managed vs. mental health managed BSS programs. Proctor model outcomes will include adoption, fidelity, penetration, and sustainability. Specific outcomes related to this framework include a) successful BSS implementation, b) fidelity in implementation of BSS, c) percentage of eligible, referred Veterans who access BSS services, and d) qualitative reports of intent to maintain the BSS program when the study is complete.

Methodology: This will be a type 2 hybrid study, combining pre- and post-implementation evaluations with a randomized clinical trial at 4 culturally diverse VA sites.

Next Steps and Implementation: Data on barriers and facilitators will be used to develop a toolkit and collaborate with study partners at the Office of Mental Health and Suicide Prevention and the National Chaplain Service to develop a national dissemination plan for BSS. The investigators will work with existing clinical staffing at the study sites, so that those sites can continue to provide BSS services after the study. Furthermore, after completing this study, BSS leaders will be qualified to train BSS leaders at other sites, creating resources for training and national dissemination.

ELIGIBILITY:
Inclusion Criteria:

Veteran status and:

* (a) validation of any of the first three items on the Moral Injury and Distress Scale, which is consistent with probable MIS
* (b) willingness to be randomized to either treatment condition
* (c) stability on mental health medications for at least 8 weeks
* (d) age of 18 years or older

Exclusion Criteria:

* (a) insufficient capacity to consent
* (b) active psychosis or substance use at levels that would interfere with treatment, assessed via chart review, the Alcohol Use Disorders Identification Test - Concise (AUDIT-C) score, and the Mini International Neuropsychiatric Interview (MINI)
* (c) currently involved in evidence-based psychotherapy for MIS, or evidence-based psychotherapy for PTSD, assessed via chart review and intake interview
* (d) managing any severe psychopathology that, in the opinion of the investigative team, requires immediate clinical attention, such as imminent suicide risk, assessed via the MINI and supplemental homicide risk questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Moral Injury and Distress Scale | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Moral Injury and Distress Scale Score Range: 0-90, with higher scores indicating more symptoms.
Change in Moral Injury Outcomes Scale | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Moral Injury and Distress Scale Score Range: 0-56, with higher scores indicating more symptoms.
Change in Expressions of Moral Injury Scale | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Expressions of Moral Injury Scale Score Range: 10-100, with higher scores indicating more symptoms.
Change in Religious and Spiritual Struggles Scale | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Religions and Spiritual Struggles Scale Score Range: 0=4 with higher scores indicating more symptoms

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Patient Health Questionnaire-9 Score range: 1-27, with higher scores indicating more symptoms
Change in Sheehan Disability Scale | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Sheehan Disability Scale Score Range: 0-30, with higher scores indicating more functional disability
Change in Inventory of Community Participation | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Inventory of Community Participation Score Range: 0-15, with higher scores indicating greater community participation
Change in Beck Scale for Suicide Ideation | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Beck Scale for Suicide Ideation Score Range: 0-38, with higher values indicating a greater risk of suicide
Change in Reasons for Living Inventory | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Reasons for Living Inventory Score Range: 48-288, with higher scores represent more reasons to live.
Change in Multiscale Measure for Postconventional Religious Functioning | 8 weeks (end of treatment) and 20 weeks (long-term follow-up)
  Full Scale Name: Multiscale Measure for Postconventional Religious Functioning. Four Subscales (Conventional Affiliate, Conventional Disaffiliate, Postconventional Affiliate, Postconventional Disaffiliate), each with a range of 12-48. Higher scores indicate religious functioning consistent with that subscale.
Client Satisfaction Questionnaire-8 | 8 weeks (end of treatment)
  Full Scale Name: Client Satisfaction Questionnaire-8 Score Range 8-32, with higher numbers indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Irene Harris, PhD MS MS, Principal Investigator — Maine VA Medical Center, Augusta, ME
Locations (5):
- United States (5):
  - Central Arkansas Veterans Healthcare System , Little Rock, AR, Little Rock, Arkansas
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Maine VA Medical Center, Augusta, ME, Augusta, Maine
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Sites involved in this study may share IPD via a) secure, VA approved videoconferencing, b) telephone, c) secure, VA approved electronic data sharing, and d) encrypted e-mail.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Study protocols will be shared across all sites in preparation for data collection across sites; individual sites will not be permitted to collect any data until they have met with lead site personnel in Maine for instruction and review of study procedures.
  The independent evaluator will be located in Maine; other sites will be expected to transmit IPD for participants scheduled for assessments within the 14 days preceding anticipated date of assessment. Data analysis will take place in Little Rock. When data collected at each individual site is complete for each Aim, the site will transmit their data to the lead statistician in Little Rock. The lead statistician may or may not transmit part or all of the data to the assistant statistician in Maine for assistance with the analysis.
Access Criteria: Only the study team will have access to this data during the study. Should the investigators receive a request for access to the data after the completion of the study, the investigators will consult with the IRB and the Privacy Officer, and if approved, share a de-identified data set as needed for verification of the research.